CLINICAL TRIAL: NCT06492551
Title: Prospective Clinical Trial of Trak Tool Usage in Post-COVID-19 Patients.
Brief Title: Post-COVID-19 Patients With Trak Tool
Acronym: TRAK-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trak Health Solutions S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PS2022011
Record Dates: First submitted 2024-07-04; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Post COVID-19 Condition
Keywords: telemedicine; COVID-19; digital health; telerehabilitation; physiotherapy; exercise program
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Exercise protocol to be performed through Trak. Trak is a rehabilitation tool and, therefore, the product of investigation.
  Interventions: Other: Trak exercise prescription protocol
- Control Group (Active Comparator): Exercise protocol with conventional methods in the Asunción Klinika gym.
  Interventions: Other: Conventional rehabilitation plan in the gym

INTERVENTIONS:
Other: Trak exercise prescription protocol — Online treatment based on therapeutic exercise using the Trak software. The patient will undergo 6 weeks of an exercise prescription protocol based on strength, balance, proprioception, and aerobic exercises. Physical therapy techniques to improve secretion management and respiratory mechanics will also be included.
  Arms: Experimental group
Other: Conventional rehabilitation plan in the gym — Treatment is based on therapeutic exercise following a conventional rehabilitation plan. The patient will undergo 6 weeks of an exercise prescription protocol based on strength, balance, proprioception, and aerobic exercises. Physical therapy techniques will also be included to improve secretion management and respiratory mechanics.
  Arms: Control Group

SUMMARY:
The clinical trial aims to analyse the effectiveness of a physiotherapeutic exercise program delivered through the telerehabilitation tool (Trak) compared to a booklet-based rehabilitation format in post-COVID-19 patients.

This research seeks to provide insights into the acceptance of the TRAK tool in this specific population, contributing to the advancement of understanding in this field.

Participants will be assigned to either the control group, which will receive conventional rehabilitation, or the experimental group, which will undergo telerehabilitation. Both groups will undergo a 6-week physical intervention, with pre- and post-intervention evaluations.

Researchers will compare the control and experimental groups to determine if there are significant differences in the health conditions of each group.

DETAILED DESCRIPTION:
The study recruitment process targets individuals who have experienced COVID-19 (moderate or severe), regardless of whether they required hospital admission, and who necessitate rehabilitation post-disease and have been discharged from quarantine.

After initial screening, individuals meeting predefined inclusion criteria will be invited to participate. Before enrollment, written informed consent will be obtained from all participants to ensure ethical compliance and respect for individual autonomy.

The primary evaluation variable selected for the study is functional capacity. Additionally, secondary assessments will include measurements of muscle strength, subjective perception of exertion, heart rate, oxygen saturation, lung capacity, and adherence to treatment (only in the experimental group).

The study cohort will comprise patients randomly assigned to experimental or control groups.

Only patients in the experimental group will receive an email containing access to the TRAK platform as part of the informed consent process. Here, they will conduct their treatment. Initial and final assessments will be performed using a digital Case Report Form for the control and experimental groups.

A rehabilitation doctor will determine the exercise protocol prescribed to the patient, which physiotherapists will administer via TRAK (experimental group) or in-person format (control group).

Patients in the experimental group will use TRAK six weeks for rehabilitation, following a prescribed exercise protocol prepared by a rehabilitation doctor. Conversely, individuals in the control group will adhere to instructions and guidelines provided by healthcare personnel during the same duration.

The study will employ an intention-to-treat analysis approach, incorporating all participants into the final analysis, regardless of their adherence to the intervention protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have suffered COVID-19 [COVID-19-moderate: clinical signs of pneumonia (fever, cough, dyspnea, tachypnea), but without signs of severe pneumonia, particularly oxygen saturation greater than or equal to 90% with air atmosphere; COVID-19-severe: clinical signs of pneumonia (fever, cough, dyspnea, tachypnea) plus one of the following: frequency respiratory > 30 inspirations/min; severe dyspnea; treatment oral medication.]
* Patients with COVID-19-related muscle pain.
* Patients with a personal device such as a tablet, smartphone, or laptop operate agilely with these devices.
* Patients with email.
* Signing of the informed consent.

Exclusion Criteria:

* Patients with a resting heart rate higher than 110 beats per minute.
* Patients with blood pressure less than 90/60 or over 160/95.
* Patients with lower blood oxygen saturation of 90%.
* Patients with advanced cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Barthel index | Baseline; up to 6 weeks
  It assesses daily activities in patients with musculoskeletal or neuromuscular conditions.

SECONDARY OUTCOMES:
Resting heart rate | Baseline; up to 6 weeks
  It is the number of times the heart beats per minute at rest, which can be an important sign of heart health.
Lung capacity | Baseline; up to 6 weeks
  It is measured by spirometry. It measures the volume of air exhaled at specific time points during complete exhalation by force, which is preceded by a maximal inhalation.
Oxygen saturation | Baseline; up to 6 weeks
  A measure of how much haemoglobin is currently bound to oxygen compared to how much is not. It is measured with a finger pulse oximeter.
Borg scale | Baseline; up to 6 weeks
  Numerical scale that ranges from 6 to 20, where 6 means "no exertion at all" and 20 means "maximal exertion".
Daniels scale | Baseline; up to 6 weeks
  It measures the patient's strength in a specific movement and muscle from 0 to 5, with 0 indicating total paralysis and 5 indicating the entire joint movement with resistance.
Trak satisfaction questionnaire | Up to 6 weeks
  The Trak satisfaction questionnaire, which was provided to patients in Spanish, consists of 12 questions about usability, usefulness, and satisfaction, as well as a suggestions section at the end.

CONTACTS AND LOCATIONS:
Overall Officials: María A García Velázquez, Principal Investigator — Asunción Klinika
Locations (1):
- Asunción Klinika, Tolosa, Gipuzkoa, Spain

REFERENCES:
- [Background] Lahham A, McDonald CF, Moore R, Cox NS, Rawlings S, Nichols A, Liacos A, Holland AE. The impact of home-based pulmonary rehabilitation on people with mild chronic obstructive pulmonary disease: A randomised controlled trial. Clin Respir J. 2020 Apr;14(4):335-344. doi: 10.1111/crj.13138. Epub 2020 Jan 11. PMID 31880078
- [Background] Zhao HM, Xie YX, Wang C; Chinese Association of Rehabilitation Medicine; Respiratory Rehabilitation Committee of Chinese Association of Rehabilitation Medicine; Cardiopulmonary Rehabilitation Group of Chinese Society of Physical Medicine and Rehabilitation. Recommendations for respiratory rehabilitation in adults with coronavirus disease 2019. Chin Med J (Engl). 2020 Jul;133(13):1595-1602. doi: 10.1097/CM9.0000000000000848. No abstract available. PMID 32251002
- [Background] Vitacca M, Malovini A, Balbi B, Aliani M, Cirio S, Spanevello A, Fracchia C, Maniscalco M, Corica G, Ambrosino N, Paneroni M. Minimal Clinically Important Difference in Barthel Index Dyspnea in Patients with COPD. Int J Chron Obstruct Pulmon Dis. 2020 Oct 21;15:2591-2599. doi: 10.2147/COPD.S266243. eCollection 2020. PMID 33116476
- [Background] Thomas P, Baldwin C, Bissett B, Boden I, Gosselink R, Granger CL, Hodgson C, Jones AY, Kho ME, Moses R, Ntoumenopoulos G, Parry SM, Patman S, van der Lee L. Physiotherapy management for COVID-19 in the acute hospital setting: clinical practice recommendations. J Physiother. 2020 Apr;66(2):73-82. doi: 10.1016/j.jphys.2020.03.011. Epub 2020 Mar 30. PMID 32312646
- [Background] Cascella M, Rajnik M, Aleem A, Dulebohn SC, Di Napoli R. Features, Evaluation, and Treatment of Coronavirus (COVID-19). 2023 Aug 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554776/ PMID 32150360